CLINICAL TRIAL: NCT06575049
Title: Comparative Analysis of Seroma and Hematoma Rates: MAXIGESIC vs. Ketorolac in Breast Cancer Surgery Patients
Brief Title: Seroma and Hematoma Rates: MAXIGESIC IV vs. Ketorolac in Breast Cancer Surgery
Status: Not yet recruiting | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hyeong-Gon Moon, PF., Seoul National University Hospital
Other Study IDs: 2312-168-1498
Record Dates: First submitted 2024-08-26; First posted 2024-08-28 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Breast Cancer; Post-Operative Hematoma; Seroma as Procedural Complication; Post-Op Complication
MeSH Terms: conditions — Breast Neoplasms; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MAXIGESIC: Maxigesig group
- Ketololac: ketololac group

SUMMARY:
The investigators aim to compare the incidence rates of seroma (fluid collection) and hematoma (blood clot) following breast cancer surgery between the conventional non-steroidal anti-inflammatory drug (NSAID) Ketorolac and MAXIGESIC. The investigators seek to determine the complication rates in patients receiving MAXIGESIC post-surgery, hypothesizing that the higher dosage of ibuprofen in MAXIGESIC compared to Ketorolac will result in lower complication rates.

ELIGIBILITY:
Inclusion Criteria:

* Systemic performance status 0-2 according to ECOG criteria
* Patients with adequate renal function: serum Cr 1.4 mg/dL or less
* Patients with adequate liver function Bilirubin, AST/ALT: 1.5 times or less of the upper limit of normal, Alkaline phosphatase: 1.8 times or less of the upper limit of normal
* Patients undergoing total mastectomy with SLNB or ALND (mastectomy and axillary sentinel lymph node dissection)
* Patients undergoing breast-conserving surgery with ALND (mastectomy and axillary dissection)
* Patients who voluntarily decided to participate in this study and signed a written informed consent form

Exclusion Criteria:

* Patients undergoing immediate reconstruction operation
* Patients with drug allergies to painkillers and anti-inflammatory drugs
* Patients with a physical condition that would interfere with understanding and submitting the consent form

Ages: 20 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Among patients who underwent breast cancer surgery at Seoul National University Hospital from January 1, 2023 to December 31, 2023, 127 patients were prescribed ketorolac and wore compression dressings. The number of patients was calculated to be approximately 60 to collect basic data to confirm the feasibility of conducting the main study.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-02-20 (Estimated)

PRIMARY OUTCOMES:
Postoperative hemovac or JP total drainage amount | within 3 months
  Postoperative hemovac or JP total drainage amount
hematoma incidence | within 3 months
  hematoma incidence
Seroma incidence | within 3 months
  Seroma incidence

SECONDARY OUTCOMES:
Length of hospital stay | within 3 months
  Length of hospital stay and re operation rate
Complication | within 3 months
  * When hematoma occurs: Whether transfusion is required and whether EB band is applied, check the amount when aspirating (diagnosis criteria color: sanguinous, old bloody [brownish], operation (hematoma evacuation)
  * When seroma occurs: check the amount when aspirating (diagnosis criteria color: serous, serosanguinous)
  * Complication: Whether abscess occurs